CLINICAL TRIAL: NCT06016933
Title: Effect of Locally Delivered Spirulina Gel on Treatment of Stage II, Grade B Periodontitis
Brief Title: Effect of Spirulina on Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Enas Elgendy, Prof. of Oral Medicine and Periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral hygiene instructions and SRP of all teeth plus placebo gel. (Placebo Comparator)
  Interventions: Procedure: SRP of all teeth
- oral hygiene instructions and SRP of all teeth, followed by insertion of the spirulina gel. (Active Comparator)
  Interventions: Drug: spirulina gel; Procedure: SRP of all teeth

INTERVENTIONS:
Drug: spirulina gel — Patient were received spirulina gel in diseased sites. The process will be repeated at 7, 14, 21 days.
  Arms: oral hygiene instructions and SRP of all teeth, followed by insertion of the spirulina gel.
Procedure: SRP of all teeth — Patients received oral hygiene instructions and SRP of all teeth.

SUMMARY:
The purpose of this study is to assess the clinical and immunological effect of spirulina in treatment of stage II periodontitis.

DETAILED DESCRIPTION:
In this study, the investigators tested the effect of spirulina gel as adjunctive of scaling and root planing in treatment of stage II, grade B periodontitis in term of probing pocket depth reduction, mean gain in clinical attachment level, and level of interleukin 6.

ELIGIBILITY:
Inclusion Criteria:

* All the patients suffer from stage II, grade B periodonitis with attachment loss 3-4 mm and probing pocket depth ≤ 5mm.

Exclusion Criteria:

* Any systemic disease that affects the periodontium. ·
* Pregnant, postmenopausal women. ·
* People who take anti-inflammatory drugs, antibiotics, or vitamins within the previous 3 month.
* People who use mouth washes regularly ·
* Participation in other clinical trials.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level | 3 months
  Clinical attachment level was measured at baseline, 1 and 3 months after gel application.
Probing pocket depth | 3 months
  Probing pocket depth was measured at baseline, 1 and 3 months after gel application.
Interleukin 6. | 3 months
  Enzyme linked immune-assay for the quantitative measurement of interleukin 6 concentration in gingival cervicular fluid at baseline, 1 and 3 months after gel application.

SECONDARY OUTCOMES:
Plaque Index | 3 months
  Plaque index was measured at baseline and at 1, and 3-months post treatment.
Gingival index | 3 months
  Gingival index was measured at baseline and at 1, and 3-months post treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided